CLINICAL TRIAL: NCT00353652
Title: Neural Mechanisms of Thiazide-induced Insulin Resistance
Brief Title: Effects of Thiazide Diuretics on Sympathetic Nervous System in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, M.D., University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 413; R01HL078782-02 (NIH)
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
Keywords: Blood Pressure, High
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Masking Description: Capsule was made to appear identical in appearance so that subjects are blinded to treatment assigned.
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Study#1: chlorthalidone (CTD) first then spironolactone (SP) (Active Comparator): Participants in study #1 only received 2 interventions. All subjects are randomized to receive 3 months of chlorthalidone first (12.5-25 mg/d), using a single-blind 2-phase crossover design. Then, the subject is transitioned to treatment with spironolactone (25-75 mg/d)without washout period for 3 months. Following 3 month treatment period, the procedures listed below were performed. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study#1: chlorthalidone (CTD), titrated dose; Drug: Study #1: spironolactone (SP), titrated dose
- Study #1: spironolactone (SP) first, then chlorthalidone (CTD) (Active Comparator): Participants in study #1 only received 2 interventions. All subjects are randomized to receive 3 months spironolactone first (25-75 mg/d), using a single-blind 2-phase crossover design. Then, the subject is transitioned to treatment with chlorthalidone(12.5-25 mg/d) without washout period. Following 3 month treatment period, the procedures listed below were performed. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study#1: chlorthalidone (CTD), titrated dose; Drug: Study #1: spironolactone (SP), titrated dose
- Study# 2 CTD alone 1st, CTD+ SP 2nd, CTD+IR 3rd (Active Comparator): Subjects are randomized to receive 3 months of fixed-dose chlorthalidone (CTD, 25 mg/d) alone first, using a single-blind 3-phase crossover design. Then, subjects are treated with fixed-dose CTD (25 mg/d) plus fixed-dosespironolactone (SP) 25 mg daily for 3 months, then fixed-dose CTD (25 mg/d) plus fixed-dose irbsesartan (IR, 150 mg daily) for 3 months. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study# 2 chlorthalidone (CTD), fixed dose; Drug: Study# 2 spironolactone (SP), fixed dose; Drug: Study# 2 irbsesartan (IR), fixed dose
- Study# 2 CTD alone 1st, CTD+IR 2nd, CTD+SP3rd (Active Comparator): Subjects are randomized to receive 3 months of fixed-dose chlorthalidone (CTD, 25 mg/d) alone first, using a single-blind 3-phase crossover design. Then, subjects are treated with fixed-dose CTD 25 mg/d plus fixed-dose irbsesartan (IR, 150 mg daily) for 3 months, followed by fixed-dose CTD (25 mg/d) plus fixed-dose spironolactone (SP) 25 mg daily for 3 months. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study# 2 chlorthalidone (CTD), fixed dose; Drug: Study# 2 spironolactone (SP), fixed dose; Drug: Study# 2 irbsesartan (IR), fixed dose
- Study# 2 CTD+SP1st, CTD alone 2nd, CTD+IR 3rd (Active Comparator): Subjects are randomized to receive fixed-dose CTD (25 mg/d) plus fixed-dose spironolactone (SP) 25 mg daily for 3 months, using a single-blind 3-phase crossover design. Then, subjects are treated with fixed-dose CTD 25 mg/d alone for 3 months, then fixed-dose CTD 25 mg/d plus fixed-dose irbsesartan (IR, 150 mg daily) for 3 months. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study# 2 chlorthalidone (CTD), fixed dose; Drug: Study# 2 spironolactone (SP), fixed dose; Drug: Study# 2 irbsesartan (IR), fixed dose
- Study# 2 CTD+SP1st, CTD+IR 2nd, CTD alone 3rd (Active Comparator): Subjects are randomized to receive fixed-dose CTD (25 mg/d) plus fixed-dose spironolactone (SP) 25 mg daily for 3 months, using a single-blind 3-phase crossover design. Then, subjects are treated with fixed-dose CTD 25 mg/d plus fixed-dose irbsesartan (IR, 150 mg daily) for 3 months, then fixed-dose CTD 25 mg/d alone for 3 months. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study# 2 chlorthalidone (CTD), fixed dose; Drug: Study# 2 spironolactone (SP), fixed dose; Drug: Study# 2 irbsesartan (IR), fixed dose
- Study# 2 CTD+IR 1st, CTD alone 2nd, CTD+SP 3rd (Active Comparator): Subjects are randomized to receive fixed-dose CTD 25 mg/d plus fixed-dose irbsesartan (IR, 150 mg daily) for 3 months, using a single-blind 3-phase crossover design. Then, subjects are treated with fixed-dose CTD 25 mg/d alone for 3 months, then fixed-dose CTD (25 mg/d) plus fixed-dose spironolactone (SP) 25 mg daily for 3 months. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study# 2 chlorthalidone (CTD), fixed dose; Drug: Study# 2 spironolactone (SP), fixed dose; Drug: Study# 2 irbsesartan (IR), fixed dose
- Study# 2 CTD+IR 1st, CTD+SP 2nd, CTD alone 3rd (Active Comparator): Subjects are randomized to receive fixed-dose CTD 25 mg/d plus fixed-dose irbsesartan (IR, 150 mg daily) for 3 months, using a single-blind 3-phase crossover design. Then, subjects are treated with fixed-dose CTD (25 mg/d) plus fixed-dose spironolactone (SP) 25 mg daily for 3 months, followed by fixed-dose CTD 25 mg/d alone for 3 months. After completion of the study procedures, the medication is discontinued.
  Interventions: Drug: Study# 2 chlorthalidone (CTD), fixed dose; Drug: Study# 2 spironolactone (SP), fixed dose; Drug: Study# 2 irbsesartan (IR), fixed dose

INTERVENTIONS:
Drug: Study#1: chlorthalidone (CTD), titrated dose — Participants in study #1 will receive 3 months of chlorthalidone (12.5-25 mg/d) at the dose titrated to achieve 24-h ambulatory BP < 130/80 mmHg
  Arms: Study #1: spironolactone (SP) first, then chlorthalidone (CTD); Study#1: chlorthalidone (CTD) first then spironolactone (SP)
Drug: Study #1: spironolactone (SP), titrated dose — Participants in study #1 will receive 3 months spironolactone (25-75 mg/d), at the dose titrated to achieve 24-h ambulatory BP < 130/80 mmHg.
  Arms: Study #1: spironolactone (SP) first, then chlorthalidone (CTD); Study#1: chlorthalidone (CTD) first then spironolactone (SP)
Drug: Study# 2 chlorthalidone (CTD), fixed dose — Participants in study #2 will receive 3 months of fixed-dose of CTD, at 25 mg/d.
  Arms: Study# 2 CTD alone 1st, CTD+ SP 2nd, CTD+IR 3rd; Study# 2 CTD alone 1st, CTD+IR 2nd, CTD+SP3rd; Study# 2 CTD+IR 1st, CTD alone 2nd, CTD+SP 3rd; Study# 2 CTD+IR 1st, CTD+SP 2nd, CTD alone 3rd; Study# 2 CTD+SP1st, CTD alone 2nd, CTD+IR 3rd; Study# 2 CTD+SP1st, CTD+IR 2nd, CTD alone 3rd
Drug: Study# 2 spironolactone (SP), fixed dose — Participants in study #2 will receive 3 months of fixed-dose SP at 25 mg daily.
  Arms: Study# 2 CTD alone 1st, CTD+ SP 2nd, CTD+IR 3rd; Study# 2 CTD alone 1st, CTD+IR 2nd, CTD+SP3rd; Study# 2 CTD+IR 1st, CTD alone 2nd, CTD+SP 3rd; Study# 2 CTD+IR 1st, CTD+SP 2nd, CTD alone 3rd; Study# 2 CTD+SP1st, CTD alone 2nd, CTD+IR 3rd; Study# 2 CTD+SP1st, CTD+IR 2nd, CTD alone 3rd
Drug: Study# 2 irbsesartan (IR), fixed dose — Participants in study #2 will receive 3 months of fixed-dose IR at150 mg daily.
  Arms: Study# 2 CTD alone 1st, CTD+ SP 2nd, CTD+IR 3rd; Study# 2 CTD alone 1st, CTD+IR 2nd, CTD+SP3rd; Study# 2 CTD+IR 1st, CTD alone 2nd, CTD+SP 3rd; Study# 2 CTD+IR 1st, CTD+SP 2nd, CTD alone 3rd; Study# 2 CTD+SP1st, CTD alone 2nd, CTD+IR 3rd; Study# 2 CTD+SP1st, CTD+IR 2nd, CTD alone 3rd

SUMMARY:
Thiazide medications are often prescribed for individuals with high blood pressure, but research has shown that they may increase an individual's risk of developing diabetes. While it is unknown exactly how thiazide causes this response, it is likely that the nervous system is somehow involved. This study will evaluate the role of the nervous system in sugar metabolism, as well as determine the effect of thiazide and other medications on individuals with high blood pressure.

DETAILED DESCRIPTION:
Thiazide medications, including chlorthalidone, are commonly prescribed for individuals with high blood pressure because they are inexpensive, effective at lowering blood pressure, and able to reduce the risk of heart failure and stroke. Despite these advantages, research has shown that thiazide medications may increase an individual's risk of developing diabetes. The exact mechanism that causes this remains unknown. Thiazide appears to increase sympathetic nervous system activity, thereby decreasing glucose reuptake and metabolism by skeletal muscle tissues. In turn, this tends to contribute to glucose intolerance and the development of diabetes. More research, however, is needed to confirm this link. Spironolactone, another blood pressure medication, does not pose the same risk for developing diabetes and may prove beneficial as a primary treatment for high blood pressure. The purpose of this study is to determine the role of the sympathetic nervous system in glucose metabolism in individuals with high blood pressure, as well as compare the effectiveness of thiazide, spironolactone, and other antihypertensive medications in reducing blood pressure. Results from this study may initiate the development of future clinical trials involving spironolactone as a primary treatment for reducing blood pressure.

This study will enroll individuals with high blood pressure. Study# 1: All subjects were randomized to receive 3 months chlorthalidone (12.5-25 mg/d) or spironolactone (50-75 mg/d), using a single-blind 2-phase crossover design without washout between treatments. Each subject was followed every 4 wk for measurement of 24-h ambulatory BP and serum potassium (K). The doses of chlorthalidone and spironolactone were titrated to achieve 24-h ambulatory BP of less than 130/80mmHg in the same subject. During chlorthalidone treatment period, subject was given oral K supplementation according to a sliding scale to maintain serum K from 4.0-4.5 mmol/liter. Then, sympathetic nerve activity (SNA) is measured after 3 months of chlorthalidone and after 3 months of spironolactone. Arterial baroreflex sensitivity, glucose, and insulin are measured at baseline, after 3 months of chlorthalidone, and after 3 months of spironolactone. Insulin sensitivity will be measured using HOMA-IR. Study #2: All subjects are randomized to 3 months of fixed-dose Chlorthalidone 25 mg once daily alone, fixed-dose Chlorthalidone 25 mg once daily plus fixed-dose Spironolactone 25 mg once daily, and fixed-dose Chlorthalidone 25 mg once daily plus fixed-dose Irbesartan 150 mg once daily, using a single-blind 3-phase crossover design without washout between treatments. Then, SNA , Arterial baroreflex sensitivity, glucose, and insulin are measured after 3 months of each treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Untreated stage 1 primary hypertension (systolic blood pressure between 140 to 159 mm Hg and diastolic blood pressure between 90 to 99 mm Hg)

Exclusion Criteria:

* Cardiopulmonary disease, as determined by medical history or by physical examination
* Serum creatinine greater than or equal to 1.5 mg/dL
* Diabetes mellitus or other systemic illness
* Left ventricular hypertrophy by echocardiography or ECG
* Hypersensitivity to chlorthalidone, spironolactone, eplerenone, angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blocker, insulin, Evans blue dye, or clonidine
* History of substance abuse (other than tobacco)
* History of gouty arthritis
* History of ACE inhibitor-induced cough or angioedema
* Evidence of secondary hypertension
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2005-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Raheja P, Price A, Wang Z, Arbique D, Adams-Huet B, Auchus RJ, Vongpatanasin W. Spironolactone prevents chlorthalidone-induced sympathetic activation and insulin resistance in hypertensive patients. Hypertension. 2012 Aug;60(2):319-25. doi: 10.1161/HYPERTENSIONAHA.112.194787. Epub 2012 Jun 25. PMID 22733474
- [Derived] Kontak AC, Wang Z, Arbique D, Adams-Huet B, Auchus RJ, Nesbitt SD, Victor RG, Vongpatanasin W. Reversible sympathetic overactivity in hypertensive patients with primary aldosteronism. J Clin Endocrinol Metab. 2010 Oct;95(10):4756-61. doi: 10.1210/jc.2010-0823. Epub 2010 Jul 21. PMID 20660053

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 119 subjects failed screening. 30 patients undergo 2-phase crossover study (chlorthalidone vs. spironolactone). 7 patients dropped out, 23 subjects completed study#1. 17 subjects undergo 3-phase study (chlorthalidone+placebo, chlorthalidone+spironolactone, and chlorthalidone+ irbesartan). 1 patients dropped out. 16 subjects completed study#2.
Period: First Intervention - 3 Months
Arm/Group | Study#1: Chlorthalidone (CTD) First Then Spironolactone (SP) | Study #1: Spironolactone (SP) First, Then Chlorthalidone (CTD) | Study# 2 CTD Alone 1st, CTD+ SP 2nd, CTD+IR 3rd | Study# 2 CTD Alone 1st, CTD+IR 2nd, CTD+SP3rd | Study# 2 CTD+SP1st, CTD Alone 2nd, CTD+IR 3rd | Study# 2 CTD+SP1st, CTD+IR 2nd, CTD Alone 3rd | Study# 2 CTD+IR 1st, CTD Alone 2nd, CTD+SP 3rd | Study# 2 CTD+IR 1st, CTD+SP 2nd, CTD Alone 3rd
Started | 15 | 15 | 6 | 7 | 3 | 0 | 1 | 0
Completed | 12 | 11 | 6 | 7 | 3 | 0 | 1 | 0
Not Completed | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention - 3 Months
Arm/Group | Study#1: Chlorthalidone (CTD) First Then Spironolactone (SP) | Study #1: Spironolactone (SP) First, Then Chlorthalidone (CTD) | Study# 2 CTD Alone 1st, CTD+ SP 2nd, CTD+IR 3rd | Study# 2 CTD Alone 1st, CTD+IR 2nd, CTD+SP3rd | Study# 2 CTD+SP1st, CTD Alone 2nd, CTD+IR 3rd | Study# 2 CTD+SP1st, CTD+IR 2nd, CTD Alone 3rd | Study# 2 CTD+IR 1st, CTD Alone 2nd, CTD+SP 3rd | Study# 2 CTD+IR 1st, CTD+SP 2nd, CTD Alone 3rd
Started | 12 | 11 | 6 | 7 | 3 | 0 | 1 | 0
Completed | 12 | 11 | 6 | 7 | 3 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention - 3 Months
Arm/Group | Study#1: Chlorthalidone (CTD) First Then Spironolactone (SP) | Study #1: Spironolactone (SP) First, Then Chlorthalidone (CTD) | Study# 2 CTD Alone 1st, CTD+ SP 2nd, CTD+IR 3rd | Study# 2 CTD Alone 1st, CTD+IR 2nd, CTD+SP3rd | Study# 2 CTD+SP1st, CTD Alone 2nd, CTD+IR 3rd | Study# 2 CTD+SP1st, CTD+IR 2nd, CTD Alone 3rd | Study# 2 CTD+IR 1st, CTD Alone 2nd, CTD+SP 3rd | Study# 2 CTD+IR 1st, CTD+SP 2nd, CTD Alone 3rd
Started | 0 | 0 | 6 | 7 | 3 | 0 | 1 | 0
Completed | 0 | 0 | 6 | 6 | 3 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 30 subjects enrolled in study#1 and 17 enrolled in study#2
Groups:
- Participants Study#1: study #1 has 2 arms. Arm 1. chlorthalidone (CTD) first then spironolactone (SP): subjects are randomized to receive 3 months of CTD first (12.5-25 mg/d), titrated to achieve 24-h BP < 130/80 mmHg. Then, the subject is transitioned to treatment with spironolactone (25-75 mg/d) without washout period for 3 months. Following 3 month treatment period, sympathetic nerve activity, 24 h-ambulatory BP, fasting plasma glucose, insulin, HOMA IR, and baroreflex sensitivity are measured. After completion of the study procedures, the medication is discontinued.
  Arm 2. spironolactone (SP) first, then chlorthalidone (CTD): subjects are randomized to receive 3 months spironolactone first (25-75 mg/d), titrated to achieve 24-h BP < 130/80 mmHg. Then, the subject is switched to CTD (12.5-25 mg/d) without washout period. Following 3 month treatment period, sympathetic nerve activity, 24 h-ambulatory BP, fasting plasma glucose, insulin, HOMA IR, and baroreflex sensitivity are measured.
- Participants Study#2: study #2 has 6 arms. Arm 1. CTD alone 1st, CTD+ SP 2nd, CTD+IR 3rd: Subjects are randomized to receive 3 months of fixed-dose chlorthalidone (CTD, 25 mg/d) alone first, using a single-blind 3-phase crossover design. Then, subjects are treated with fixed-dose CTD (25 mg/d) plus fixed-dosespironolactone (SP) 25 mg daily for 3 months, then fixed-dose CTD (25 mg/d) plus fixed-dose irbsesartan (IR, 150 mg daily) for 3 months.
  Arm 2. fixed-dose CTD alone 1st, CTD+IR 2nd, CTD+SP3rd Arm3. fixed-dose CTD+SP1st, CTD alone 2nd, CTD+IR 3rd Arm 4. fixed-dose CTD+SP1st, CTD+IR 2nd, CTD alone 3rd Arm 5. CTD+IR 1st, CTD alone 2nd, CTD+SP 3rd Arm 6. CTD+IR 1st, CTD+SP 2nd, CTD alone 3rd
- Total: Total of all reporting groups
Arm/Group | Participants Study#1 | Participants Study#2 | Total
Number analyzed (Participants) | 30 | 17 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (2.0) | 50.6 (2.3) | 49.7 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 21 | 13 | 34
Region of Enrollment [Number; unit: participants]
  United States | 30 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Sympathetic Nerve Activity
Time Frame: Measured at 3 months
Measure: Mean (Standard Error); unit: bursts/min
Groups:
- Study#1: Chlorthalidone (CTD), Titrated Dose: Participants in study #1 only received 2 interventions. All subjects are randomized to receive 3 months of chlorthalidone first (12.5-25 mg/d) or spironolactone (25-75 mg/d) first at the dose titrated to achieve 24-h ambulatory BP < 130/80 mmHg, using a single-blind 2-phase crossover design. Then, the subject is transitioned to treatment the remain arm without washout period for 3 months. Following 3 month treatment period, measurement of outcomes are performed. After completion of the study procedures, the medication is discontinued.
- Study #1: Spironolactone (SP), Titrated Dose: Participants in study #1 only received 2 interventions. All subjects are randomized to receive 3 months of spironolactone (25-75 mg/d) first or chlorthalidone first (12.5-25 mg/d) at the dose titrated to achieve 24-h ambulatory BP < 130/80 mmHg, using a single-blind 2-phase crossover design. Then, the subject is transitioned to treatment the remain arm without washout period for 3 months. Following 3 month treatment period, measurement of outcomes are performed. After completion of the study procedures, the medication is discontinued.
- Study# 2 Chlorthalidone (CTD), Fixed Dose; Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose; Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose: Subjects are randomized to receive 3 months of fixed-dose chlorthalidone (CTD, 25 mg/d) alone first or fixed-dose CTD (25 mg/d) plus fixed-dose spironolactone (SP) 25 mg daily first or fixed-dose CTD (25 mg/d) plus fixed-dose irbsesartan (IR, 150 mg daily) first, using a single-blind 3-phase crossover design. Then, subjects are treated with the remaining one of the 2 arms for 3 months, followed by the last arm for 3 months without washout period. After completion of the study procedures, the medication is discontinued.
Arm/Group | Study#1: Chlorthalidone (CTD), Titrated Dose | Study #1: Spironolactone (SP), Titrated Dose | Study# 2 Chlorthalidone (CTD), Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose
Number analyzed (Participants) | 23 | 23 | 17 | 17 | 17
bursts/min | 46 (4) | 40 (3) | 49 (3) | 42 (3) | 52 (2)

2. Secondary Outcome: 24-hour Ambulatory Systolic Blood Pressure
Time Frame: Measured at 3 months
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Study #1: Spironolactone (SP), Titrated Dose: Participants in study #1 only received 2 interventions. All subjects are randomized to receive 3 months of chlorthalidone first (12.5-25 mg/d) or spironolactone (25-75 mg/d) first at the dose titrated to achieve 24-h ambulatory BP < 130/80 mmHg, using a single-blind 2-phase crossover design. Then, the subject is transitioned to treatment the remain arm without washout period for 3 months. Following 3 month treatment period, measurement of outcomes are performed. After completion of the study procedures, the medication is discontinued.
Arm/Group | Study#1: Chlorthalidone (CTD), Titrated Dose | Study #1: Spironolactone (SP), Titrated Dose | Study# 2 Chlorthalidone (CTD), Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose
Number analyzed (Participants) | 23 | 23 | 17 | 17 | 17
mmHg | 127.4 (2) | 128.6 (2) | 123.5 (2) | 121.6 (3) | 119.8 (3)

3. Secondary Outcome: Insulin
Description: fasting plasma insulin
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: mU/liter
Groups:
- Study# 2 CTD Fixed Dose 25 mg/d; Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose; Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose: Subjects are randomized to receive 3 months of fixed-dose chlorthalidone (CTD, 25 mg/d) alone first or fixed-dose CTD (25 mg/d) plus fixed-dose spironolactone (SP) 25 mg daily first or fixed-dose CTD (25 mg/d) plus fixed-dose irbsesartan (IR, 150 mg daily) first, using a single-blind 3-phase crossover design. Then, subjects are treated with the remaining one of the 2 arms for 3 months, followed by the last arm for 3 months without washout period. After completion of the study procedures, the medication is discontinued.
Arm/Group | Study#1: Chlorthalidone (CTD), Titrated Dose | Study #1: Spironolactone (SP), Titrated Dose | Study# 2 CTD Fixed Dose 25 mg/d | Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose
Number analyzed (Participants) | 23 | 23 | 17 | 17 | 17
mU/liter | 8.24 [4.56 to 10.49] | 7.6 [4.68 to 8.6] | 7.6 [4.08 to 19.7] | 4.87 [3.50 to 6.78] | 6.8 [3.28 to 10.25]

4. Secondary Outcome: HOMA-IR
Description: assessment of insulin resistance calculated by multiplying fasting plasma insulin (mU/l) with fasting plasma glucose (mmol/l) divided by 22.5.
Time Frame: 3 months
Population: unequal randomization by chance
Measure: Median (Inter-Quartile Range); unit: mU/l*mmol/l
Arm/Group | Study#1: Chlorthalidone (CTD), Titrated Dose | Study #1: Spironolactone (SP), Titrated Dose | Study# 2 Chlorthalidone (CTD), Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose
Number analyzed (Participants) | 23 | 23 | 17 | 17 | 17
mU/l*mmol/l | 1.91 [1.17 to 2.96] | 1.33 [0.56 to 2.06] | 1.87 [0.8 to 4.13] | 0.85 [0.69 to 1.52] | 1.42 [0.77 to 2.23]

5. Secondary Outcome: Sympathetic Baroreflex Sensitivity
Description: slope relating percent change in SNA (% change in total activity from baseline) to diastolic BP.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: % change from baseline per mmHg
Groups:
- Drug: Study #1: Spironolactone (SP), Titrated Dose: Participants in study #1 only received 2 interventions. All subjects are randomized to receive 3 months of spironolactone (25-75 mg/d) first or chlorthalidone first (12.5-25 mg/d) at the dose titrated to achieve 24-h ambulatory BP < 130/80 mmHg, using a single-blind 2-phase crossover design. Then, the subject is transitioned to treatment the remain arm without washout period for 3 months. Following 3 month treatment period, measurement of outcomes are performed. After completion of the study procedures, the medication is discontinued.
Arm/Group | Study#1: Chlorthalidone (CTD), Titrated Dose | Drug: Study #1: Spironolactone (SP), Titrated Dose | Study# 2 Chlorthalidone (CTD), Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose
Number analyzed (Participants) | 23 | 23 | 17 | 17 | 17
% change from baseline per mmHg | -9.1 (3.8) | -15.2 (3.2) | -12.9 (7.8) | -11.3 (8.8) | -12.0 (7)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Study#1: Chlorthalidone (CTD), Titrated Dose | Study #1: Spironolactone (SP), Titrated Dose | Study# 2 Chlorthalidone (CTD), Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose | Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/26 | 0/27 | 0/17 | 0/17 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study#1: Chlorthalidone (CTD), Titrated Dose (N=26) | Study #1: Spironolactone (SP), Titrated Dose (N=27) | Study# 2 Chlorthalidone (CTD), Fixed Dose (N=17) | Study# 2 CTD Fixed Dose 25 mg/d Plus SP Fixed Dose (N=17) | Study# 2 CTD Fixed Dose 25 mg/d Plus IR Fixed Dose (N=17)
chest pain (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes